CLINICAL TRIAL: NCT00895713
Title: Efficacy and Safety of Intramuscular Hepatitis B Virus Immune Globulin Grifols for the Prevention of Hepatitis B Virus Recurrence After Orthotopic Liver Transplantation.
Brief Title: Efficacy and Safety of Intramuscular HBIG Grifols for the Prevention of Recurrence After Liver Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Antonio Páez, MD, Instituto Grifols S.A.
Organization: Grifols Biologicals, LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IG302
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-05

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B; HBV; Anti-hepatitis B antibodies; Immunoglobulins; liver transplantation; Protective levels; Recurrence; Intramuscular
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Recurrence | interventions — igantibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- im HBIG Grifols (Experimental)
  Interventions: Drug: intramuscular hepatitis B virus immune globulin

INTERVENTIONS:
Drug: intramuscular hepatitis B virus immune globulin — Biweekly intramuscular doses of 2000 IU administered during 6 consecutive months
  Other Names: Igantibe

SUMMARY:
The purpose of this study is to determine if treatment with intramuscular hepatitis B virus immune globulin Grifols, a new specific hepatitis B immune globulin, is effective and safe for the prevention of hepatitis B virus recurrence after orthotopic liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Age > 18 years and < 70 years.
3. OLT recipient for HBV infection-related disease for > 18 months before inclusion in the clinical trial.
4. Serum HBsAg-positive within 3 months before transplantation.
5. Serum HBsAg-negative just before inclusion in the clinical trial.
6. Serum HbeAg-negative just before inclusion in the clinical trial.
7. Serum HBV DNA-negative by DNA PCR-amplification assay (lower detection limit 102 genomes/ml) just before inclusion in the clinical trial.
8. Continuous and interrupted prophylaxis with HBIG after an-hepatic phase as part of the subject clinical care.
9. Trough serum HBsAg Ab (HBsAg IgG) titer (immediately pre-dose) > 150 I.U./l in at least 2 consecutive determinations within last 3 months before inclusion in the clinical trail.
10. Signed informed consent.

Exclusion Criteria:

1. Serum HBsAg-positive just before inclusion in the clinical trial.
2. Serum HBeAg-positive within 3 months before transplantation.
3. Serum HBV DNA-positive by standard DNA hybridisation assay (lower detection limit 105 genomes/ml), or by any less sensitivity technique, within 3 months before transplantation.
4. Unknown serum HBV replication status (no data about HbeAg and HBV DNA) within 3 months before transplantation.
5. Previous recurrence of HBV in the transplanted liver defined by serum HBV DNA- positive by sensitive hybridisation (lower detection limit 105 genomes/ml) assay or any less sensitive technique, and/or serum HBeAg-positive, and/or serum HBsAg-positive.
6. Re-transplanted liver even for reasons not related to HBV infection.
7. Evidence of hepatocellular carcinoma in the transplanted liver, or metastatic disease, at time of inclusion in the clinical trial.
8. Evidence of graft rejection at time of inclusion in the clinical trial.
9. Life-expectancy less than 1 year.
10. VHC infection.
11. HIV type 1 or type 2 infection.
12. Acute HAV infection.
13. Previous treatment with i.m. HBIG Grifols within 3 months before inclusion in the clinical trial.
14. Intolerance or allergy to any i.m. HBIG Grifols containing substance (glycine, sodium chloride, sterile water for injection, homologous human immune globulin).
15. History of SAEs related to the administration of human blood-derived products.
16. History of frequent AEs, even non-serious, related to the administration of human blood-derived products.
17. Selective IgA deficiency with Abs against IgA.
18. Platelet count < 50 x 109/L.
19. Prothrombin time (PT) < 60%.
20. Activated partial thromboplastin time (APTT) ratio > 1.5.
21. Any haemostatic abnormality contraindicating i.m. injection according to investigator's judgement.
22. Haemoglobin < 11 g/dl.
23. Alcohol or drug abuse at the moment or within 1 year before inclusion in the clinical trial.
24. Pregnant woman or woman who is expecting to be pregnant within 1 year after inclusion in the clinical trial.
25. Breast-feeding woman.
26. Any severe acute or chronic medical, surgical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, or may interfere with the interpretation of study results and, in the judgment of the investigator, makes the subject inappropriate for entry in this clinical trial.
27. Impossibility to donate a serum sample before the first investigational product administration.
28. Planned treatment with Ig other than i.m. HBIG Grifols within the clinical trial period.
29. Planned modification, during the clinical trial period, of the prophylactic regimen with nucleoside analogues followed by the subjects, if any, within last 3 months before inclusion in the clinical trial.
30. The subject has been previously admitted to this clinical trial.
31. Participation in other clinical trial within 3 months before study inclusion.
32. Subject's incapacity of giving consent personally.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-11; Primary Completion 2005-06 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Mean trough serum HBsAg Ab titer | Months 4-6

SECONDARY OUTCOMES:
HBV recurrence percentage in long-term OLT recipients during i.m. HBIG Grifols treatment period | Week 2 - 7 months
Mean trough HBsAg Ab titer | 4 months
Individualised trough HBsAg Ab titer | Week 2 - 7 months
Number of subjects with serum HBV DNA-positive samples by DNA PCR-amplification assay | Week 2 - 7 months
Safety and tolerability | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Franco Filipponi, Prof. MD, Principal Investigator — Liver Transplantation Co-ordinating Section. Cisanello Hospital. (University of Pisa).
Locations (2):
- Italy (2):
  - Cisanello Hospital. (University of Pisa)., Pisa
  - Ospedaliera Molinette, Torino